CLINICAL TRIAL: NCT05528978
Title: Impact of Inner Engineering Yoga Program on Interpersonal Relationships
Brief Title: Impact of Inner Engineering on Relationships
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Professor of Anesthesia, Beth Israel Deaconess Medical Center
Other Study IDs: 2022P000587
Record Dates: First submitted 2022-08-29; First posted 2022-09-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Relationship, Social
Keywords: Yoga; Stress; Wellbeing; Mindfulness; Meditation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inner Engineering Intervention: The intervention investigators propose for the study includes an Online Course with 7 modules, or a 10 hours long course, and a 1-2 day In-Person Course, in which participants will learn a simple 21 minute practice called Shambhavi Mahamudra Kriya, also known as Shambhavi Kriya.
  Interventions: Behavioral: Shambhavi Kriya

INTERVENTIONS:
Behavioral: Shambhavi Kriya — The intervention investigators propose for the study includes an Online Course with 7 modules, or a 10 hours long course, and a 1-2 day In-Person Course, in which participants will learn a simple 21 minute practice called Shambhavi Mahamudra Kriya, also known as Shambhavi Kriya.
  Shambhavi Kriya is a powerful and purifying energy technique incorporating the breath. This practice is said to align the participants system such that their body, mind and emotions function in harmony.

SUMMARY:
This study aims to assess the impact of Shambhavi Mahamudra Kriya on human relationships in terms of overall well-being associations with interpersonal and relational outcomes.

Specific aims include:

1. To quantitatively assess the impact of Shambhavi Mahamudra Kriya on measures of relationship quality, interpersonal mindfulness, and overall well-being
2. To qualitatively explore the experience and the general Social and Relational impact of Shambhavi Mahamudra Kriya on participants.

DETAILED DESCRIPTION:
This observational cross-sectional study aims to enroll participants who are already registered for an Inner Engineering program to learn Shambhavi Mahamudra Kriya

The practice participants are learning is a multi-component 21-minute meditation called Shambhavi Mahamudra Kriya. It is offered by the non-profit Isha Foundation. It incorporates a combination of different breathing patterns and meditative components. The intervention training provides precise, step by step and easy to follow instructions on how to perform this practice. Performed in a seated posture, this is a simple, safe and accessible intervention that requires no previous experience of meditation.

Some Inner Engineering programs where participants learn Shambhavi Mahamudra Kriya have a pre-requisite of taking the Inner Engineering Online (IEO) program. The IEO program consists of seven online modules. These modules give the participants an opportunity to intellectually explore the basics of life using methods that are from the distilled essence of yogic sciences. The course imparts wisdom to manage the body, mind, emotions, and the fundamental life energy within.

Importantly, the participants would be able to attend their Inner Engineering program and subsequent meditation and yoga practices would occur regardless of whether or not they decided to participate in the study.

With this study we aim to evaluate the impact of Shambhavi Kriya on relationships using validated scales and qualitative analysis. Enrollment into the study will be ongoing until we are able to get a sufficient sample size. Apart from the surveys and qualitative interviews at select points over a 6-month period, there is no additional study procedures involved in the study, details of which are discussed below.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have registered to take an Inner Engineering program to learn Shambhavi Mahamudra Kriya.
* Participants must be able to read and understand English.

Exclusion Criteria:

* Not currently residing in United States
* Below the age of 18

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This population has enrolled in an Inner Engineering program to learn Shambhavi Mahamudra Kriya.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2022-11-13 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Relationship Quality (PN-RQ) over 6 months | Data collection at baseline, immediately after the intervention, week 6, 6 months
  PN-RQ Scale is a 16-item validated instrument that assesses relationship quality. On a 7-point Likert Scale (1= not at all, 7= completely) participants rate eight different positive and negative qualities they attribute to their relationship. The average item score in each category is compared, with the higher score indicating the dominating relationship quality.

SECONDARY OUTCOMES:
Change in Perceived Stress Scale (PSS) over 6 months | Data collection at baseline, immediately after the intervention, week 6, 6 months
  PSS is a 10-question validated instrument that assesses stress. Participants are asked to rate on a scale of 0 (never) to 4 (very often) how often they agree with various statements. Items from each of the 10 questions are then summed to create a total perceived stress score. This scale will be employed as an online scale which will be utilized by participants to self-report on perceived stress for the purpose of this study.
Change in Interpersonal Mindfulness Scale (IMS) over 6 months | Data collection at baseline, immediately after the intervention, week 6, 6 months
  IMS is a 27-item validated instrument that assesses mindfulness in the context of interpersonal interactions grouped into four subscales: presence, awareness of self and others, nonjudgmental acceptance, and nonreactivity. Each statement is rated on a 5-point Likert scale (1= almost never to 5= almost always).
Change in Flourishing Scale over 6 months | Data collection at baseline, immediately after the intervention, week 6, 6 months
  The Flourishing Scale is 12-item validated instrument that assess overall well-being in 5 domains: happiness and life satisfaction, mental and physical health, meaning and purpose, character and virtue, and close social relationships. The "Flourish" measure is the sum of the scores from each of the five domains. The "Secure Flourish" measure includes the financial and material stability domain. Questions are assessed on a scale of 0-10 (0= Not satisfied at all, 10= Completely satisfied).
Compliance questionnaire | weekly for 6 weeks post-Inner Engeineering program and monthly for 6 months.
  The weekly compliance questionnaire is a tool which helps the participants to keep track of their activities each week. This enables the study team to measure compliance and protocol adherence by the participants by collecting information on their routine activity practiced, its frequency and duration.
Qualitative Interviews | Between week 6-16 weeks
  The semi-structured individual interviews will allow us to gain rich, descriptive information about the participant's experience with the Shambhavi Kriya practice, and the general impact of the practice on the participants. The semi-structured interviews will ensure a systematic and flexible approach to data collection. The interviews will cover the following main topics:
  1. Participants' experience with Shambhavi Kriya practice and
  2. Perceptions of the participants of themselves before and after completing 6 weeks of the practice.
Change in Compassion Scale (CS) over 6 months | Data collection at baseline, immediately after the intervention, week 6, 6 months
  The Compassion Scale is a 16-item validated instrument that assess an individual's level of compassion to others in four subscales: Indifference, kindness, mindfulness, and common humanity, Each statement is rated on a 5-point Likert scale (1=almost never, 5= almost always).
Change in Satisfaction Survey | At week 6 and 6 months
  This survey will collect the participants' feedback on the study and Shambhavi Mahamudra Kriya.

CONTACTS AND LOCATIONS:
Overall Officials: Balachundar Subramaniam, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Centre, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jafari N, Manvelian A, Mohamed E, Rayapuraju A, Orui H, Alkuhaimi S, Reed PU, Subramaniam B. Inner engineering is associated with perceived improvements in relationship quality, interpersonal connections, and interpersonal compassion. Front Psychol. 2024 Dec 23;15:1454293. doi: 10.3389/fpsyg.2024.1454293. eCollection 2024. PMID 39764085